CLINICAL TRIAL: NCT05558059
Title: Elucidating Perifoveal Vasculature Development in Infants
Brief Title: Imaging Retinal Vasculature in Infant Eyes
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00111105; 1R01EY03413401 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2022-09-06; First posted 2022-09-28 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; Optical Coherence Tomography; Perifoveal vasculature; Vascular development; Macular edema; ROP; OCT; Prematurity; Optical Coherence Tomography Angiography; OCTA
MeSH Terms: conditions — Retinopathy of Prematurity; Macular Edema; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: 16 preterm infants undergoing ROP screening to optimize methods to acquire and process beside infant perifoveal vascular imaging and assess rigor and reproducibility.
  The visits in the ICN (Intensive Care Nursery) will occur between 32 and 43 weeks post menstrual age at the time of ROP screening exams. Study visits will include, but are not limited to:
  * Ocular examination
  * OCT imaging of retinal microanatomy
  * OCTA imaging of retinal microvasculature
  * Medical and ocular history
  * Adverse event documentation
  Interventions: Device: Handheld Optical Coherence Tomography with OCT Angiography

INTERVENTIONS:
Device: Handheld Optical Coherence Tomography with OCT Angiography — OCT systems are in vivo optical imaging technology that allows non-contact imaging of early-stage ocular pathology. They create real-time, non-invasive images of ocular microstructure and have become standard-of-care instruments in ophthalmic imaging in clinics and operating rooms. In contrast to the visible light used in clinical eye examinations, because infrared light is not visible, the participant is not disturbed by the light. OCT imaging allows the capture of hundreds of B-scan (cross-sectional) images in seconds. These B-scans are analyzed for depth-resolved information and can also be stacked to create a volume and the stack may be summed up to create a retinal image.
  OCT angiography (OCTA) is an extension of the OCT systems, by taking images at the same location over time to extract retinal vascular flow information. It has been utilized to assess the ocular blood flow in many adult and pediatric patients.
  Other Names: Handheld OCT and OCTA

SUMMARY:
Retinopathy of prematurity is a leading cause of childhood blindness worldwide. The fovea, a critical location in the retina determining visual acuity and visual function, and the blood vessels around it, are abnormally developed in infants with retinopathy of prematurity. However, how these blood vessels form during development of the human fovea remains unclear. This research will advance our understanding of the fundamental knowledge of how the blood vessels around the fovea form in infants, and how they change in diseased states such as preterm birth or retinopathy of prematurity.

ELIGIBILITY:
Inclusion Criteria:

* Health care provider, knowledgeable of protocol, agrees that study personnel could contact the Parent/Legal guardian
* Parent/Legal Guardian is able and willing to consent to study participation for the infant
* Infant meets the American Association of Pediatrics eligibility of ROP screening, and is age less than 34 6/7 weeks postmenstrual age at first visit

Exclusion Criteria:

* Participant or Parent/Legal Guardian unwilling or unable to provide consent
* Infant has a health or eye condition that preclude eye examination or retinal imaging (e.g. corneal opacity such as with Peter's anomaly or cataract)
* Infant has a health condition, other than prematurity, that has a profound impact on brain development (e.g. anencephaly)

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants undergoing screening for retinopathy of prematurity
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in vascular density of intermediate and deep vascular plexus at the fovea and perifovea | During hospitalization (at approximately 32-44 weeks post menstrual age, PMA)
  Measured by retinal OCTA imaging.

SECONDARY OUTCOMES:
Change in vascular density of superficial vascular plexus at the fovea and perifovea | During hospitalization (at approximately 32-44 weeks post menstrual age, PMA)
  Measured by retinal OCTA imaging.
Change in avascular zone size of superficial, intermediate and deep vascular plexus | During hospitalization (at approximately 32-44 weeks post menstrual age, PMA)
  Measured by retinal OCTA imaging.
Change in network length of intermediate and deep vascular plexus | During hospitalization (at approximately 32-44 weeks post menstrual age, PMA)
  Vascular density of superficial vascular plexus at the fovea and perifovea; Avascular zone size of superficial, intermediate and deep vascular plexus; Network morphology of intermediate and deep vascular plexus; Network length of intermediate and deep vascular plexus.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Chen, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Elucidating Perifoveal Vascular Development in Infants study data cannot be analyzed for publication until they are released by the study Principal Investigator upon final review and approval by the Data Safety and Monitoring Committee.
  Data will be made available as follows:
  * A summary, de-identified data set available upon request through direct inquiries to the Study PI or Statistical Analysis Center a year after publication.
  * By the end of the funding period, de-identified SAS data sets and form images corresponding to all data collection forms, as well as key derived variables, will be put on file with a data repository.
  * Researchers may request limited access data sets.
  * The raw and analyzed imaging datasets will be made available after the completion of this study.
  Approved recipients will need to enter into a data sharing agreement. Costs for compilation and access to the datasets will be the responsibility of the recipients.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available after the completion of the study.
Access Criteria: Data requests must be submitted to the PI or the Statistical Analysis Center. Approved recipients will need to enter into a data sharing agreement.
  Costs for compilation and access to the datasets will be the responsibility of the recipients.